CLINICAL TRIAL: NCT00959140
Title: Phase II Study for Standardization of CD3+ T Cell Dose for Patients Receiving Allogeneic Peripheral Blood Stem Cell Transplants From Matched Related Donors
Brief Title: Standardization of CD3+ T Cell Dose for Patients Receiving Allogeneic Peripheral Blood Stem Cell Transplantation From Matched Related Donors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Miltenyi Biotec, Inc. (Industry)
Responsible Party: Principal Investigator, Antonio Di Stasi, Primary Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB 1410
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Allo PBSC; HSCT; Bone Marrow Transplant; Allogeneic Bone Marrow Transplant; Matched Related Donor Transplant; MRD HSCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CD3+ T-cell depletion (Experimental): CD3+ T-cell depletion
  Interventions: Device: CD3+ T cell depletion

INTERVENTIONS:
Device: CD3+ T cell depletion — The peripheral blood stem cell product is engineered to deliver a dose of 15 to 20 x10^7 CD3+ cells/kg recipient body weight. Other components of the graft will not be manipulated and the recipient will receive the total number of cells collected with the exception of minimal losses that occur during the process of CD3+ T cell isolation. Following collection, CD3+ T cells will be enumerated and a portion of the product containing 15 to 20 x10^7 CD 3+ cells/kg will be set aside. The remainder of the product will be depleted of CD3+ T cells.
  Following CD3+ T cell depletion, the CD3+ T cell depleted product will then be combined with the unmanipulated product to provide the specified levels of CD3+ T cells/kg recipient body-weight. The graft is infused into the patient on the same day as selected and within 24 hours of donor aphaeresis.

SUMMARY:
Stem cells collected from sibling donors for allogenic transplants contain various types of cells. The predominant immune cells are called CD3+ T cells. The amount of these T cells vary vastly from donor to donor. This study is to determine if standardizing the CD3+ T cell dose will benefit the recipient (patient). As well as to help discover if dose standardization causes less variation in outcomes between patients and to make transplantation more predictable and complications easier to manage.

DETAILED DESCRIPTION:
The optimal CD3+ cell dose to be used for allo HSCT is unknown. In addition, there are multiple variables in addition to CD3+ cell dose which affect engraftment, immune reconstitution, GVH and GVL in these patients including recipient age, diagnosis, disease status at transplantation, donor/recipient tissue type match, preparative regimen, and GVHD prophylaxis. Thus the ability to produce products with a fixed CD3+ content is critical to further research and ultimately to the definition of the "right dose" of CD3+ cells for various clinical situations.

Patients who meet eligibility criteria will receive a peripheral blood stem cell product from their original matched sibling donor engineered to deliver a dose of 3.0+/-0.5 x107 CD3+ cells/kg recipient body weight. Other components of the graft will not be manipulated and the recipient will receive the total number of cells collected with the exception of minimal losses that occur during the process of CD3+ T cell isolation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥19 years of age.
2. Patients must meet all the UAB diagnosis and disease status criteria for clinical appropriateness for myeloablative allo HSCT derived from ASBMT and NCCN guidelines.
3. Patients must have a 10/10 HLA matched sibling (excluding identical twin). All donors will be evaluated for eligibility and suitability per standard of care according FACT and NMDP guidelines.
4. Adequate organ function: All organ function testing should be done within 28 days of study registration.
5. Cardiac: Left ventricular ejection fraction (LVEF) ≥ 50% by MUGA (Multi Gated Acquisition) scan or echocardiogram.
6. Pulmonary: FEV1 (Forced expiratory volume in 1 second) and FVC (Forced vital capacity) ≥ 50% predicted, DLCO (alveolar diffusion capacity for carbon monoxide) (corrected for hemoglobin) ≥ 50% of predicted.
7. Renal: The estimated creatinine clearance (CrCl) must be equal or greater than 60 mL/min/1.73 m2 as calculated by the Cockcroft-Gault Formula
8. Performance status: Karnofsky ≥ 70%
9. Hepatic (values to be less than what is considered grade II toxicity per the CTCAE (common terminology criteria for adverse events)

Exclusion criteria

1. Uncontrolled infections, defined as positive blood cultures within 72 hours of study entry, or evidence of progressive infection by imaging studies such as chest CT scan within 14 days of registration.
2. HIV positive patients.
3. Prior autologous or allogeneic transplantation for any disease.
4. Scheduled to receive non-myeloablative or reduced intensity conditioning regimen.
5. High Risk Features associated with increased relapse risk or poor outcomes:

   1. AML/ALL: with Bi-phenotypic features
   2. AML: Refractory to Induction and salvage therapy
   3. ALL: Refractory to Induction and salvage therapy
   4. CML: Active blast crisis
   5. HL: Disease refractory to chemotherapy or targeted therapy
   6. NHL: Disease refractory to chemotherapy or targeted therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of acute graft versus host disease (aGVHD) with the chosen fixed dose of CD3+ cells | 1 year

SECONDARY OUTCOMES:
Time to engraftment | 60 days
State of chimerism over time | 2 years
Immune reconstitution over time | 2 years
Incidence, severity and organ involvement with chronic GVHD (cGVHD) | 2 years
Overall survival | 2 years
Disease free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Saad, MD, Principal Investigator — University of Alabama in Birmingham
Locations (1):
- University of Alabama Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMTCT Program Web Site — http://www.uab.edu/medicine/bonemarrow/